CLINICAL TRIAL: NCT05465668
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of DWP16001 Drug A and DWP16001 Drug C in Healthy Adult Volunteers
Brief Title: Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics of DWP16001 Drug A and C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001106
Record Dates: First submitted 2022-07-05; First posted 2022-07-20 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: DWP16001 Drug A (Experimental): 1 tablet, Oral, once daily single dose
  Interventions: Drug: DWP16001 Drug A
- Intervention: DWP16001 Drug C (Experimental): 1 tablet, Oral, once daily single dose
  Interventions: Drug: DWP16001 Drug C

INTERVENTIONS:
Drug: DWP16001 Drug A — DWP16001 Drug A
  Arms: Intervention: DWP16001 Drug A
Drug: DWP16001 Drug C — DWP16001 Drug C
  Arms: Intervention: DWP16001 Drug C

SUMMARY:
This study aims to evaluate the safety and pharmacokinetic characteristics after administration of DWP16001 Drug A and DWP16001 Drug C in healty adult volunteers.

DETAILED DESCRIPTION:
The study design is a Randomized, Open-label, Oral, Single-dose, Two-way crossover study. The patients were randomly assigned to each group. Primary endpoint was Cmax and AUClast of DWP16001. Secondary endpoints were AUCinf, AUClast, Tmax, t1/2, CL/F, and Vd/F of DWP16001.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with a body weight of ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 30.0 kg/m2

☞ BMI (kg/m2) = Body weight (kg) / {Height (m)}2

Exclusion Criteria:

* musculoskeletal diseases
* mental diseases
* hemato-oncologic diseases

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of DWP16001 | At pre-dose (0 hour), and post-dose 0.25 to 72 hour.
  Peak Plasma Concetration of DWP16001
AUClast of DWP16001 | At pre-dose (0 hour), and post-dose 0.25 to 72 hour.
  The area under the plasma drug concentration-time curve of DWP16001

SECONDARY OUTCOMES:
Tmax of DWP16001 | At pre-dose (0 hour), and post-dose 0.25 to 72 hour.
  Time at Cmax of DWP16001
T1/2 of DWP16001 | At pre-dose (0 hour), and post-dose 0.25 to 72 hour.
  Half life of DWP16001
CL/F of DWP16001 | At pre-dose (0 hour), and post-dose 0.25 to 72 hour.
  Apparent total clearance of the drug from plasma after oral administration of DWP16001
Vd/F of DWP16001 | At pre-dose (0 hour), and post-dose 0.25 to 72 hour.
  Volume of distribution of DWP16001

CONTACTS AND LOCATIONS:
Locations (1):
- CHA unuversity bundang medical center, Seongnam, South Korea